CLINICAL TRIAL: NCT00940485
Title: A Study on Optimizing HBeAg Seroconversion in HBeAg Positive CHB Patients With Combination or Sequential Treatment of Pegylated Interferon Alpha-2a and Entecavir
Brief Title: A Study of Combination or Sequential Treatment With PEGASYS (Peginterferon Alfa-2a) and Entecavir in Patients With HBeAg Positive Chronic Hepatitis B
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML22265
Record Dates: First submitted 2009-06-16; First posted 2009-07-16 (Estimated); Results first posted 2016-02-22 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-02

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir; peginterferon alfa-2a

ARMS (2):
- Peginterferon alfa-2a + entecavir (Experimental): Participants received PEGASYS® (peginterferon alfa-2a)180 micrograms (mcg) subcutaneously once weekly for 48 weeks, plus entecavir 0.5 milligram (mg) orally once daily for 8 weeks.
  Interventions: Drug: entecavir; Drug: peginterferon alfa-2a [Pegasys]
- Entecavir (Active Comparator): Participants received entecavir 0.5 mg orally once daily for 48 weeks.
  Interventions: Drug: entecavir

INTERVENTIONS:
Drug: entecavir — 0.5mg po daily for 8 weeks
  Arms: Peginterferon alfa-2a + entecavir
Drug: entecavir — 0.5mg po daily for 48 weeks
  Arms: Entecavir
Drug: peginterferon alfa-2a [Pegasys] — 180 micrograms sc/week for 48 weeks
  Arms: Peginterferon alfa-2a + entecavir

SUMMARY:
This 2 arm study will assess the efficacy and safety of Pegasys in combination or sequential treatment with entecavir in patients with HBeAg positive chronic hepatitis B. Patients who have been pretreated with, and responded to, entecavir for 9 to 36 months were randomized to one of 2 groups, to receive Pegasys 180micrograms/week sc for 48 weeks + entecavir 0.5mg po daily for 8 weeks, or entecavir 0.5mg po daily for 48 weeks. The anticipated time on study treatment is 3-12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >=18 and </= 65 years of age
* HBeAg positive chronic hepatitis B
* Pre-treatment with entecavir for 9-36 months

Exclusion Criteria:

* Antiviral, antineoplastic or immunomodulatory treatment
* Co-infection with active hepatitis A, C or D, or HIV
* Evidence of decompensated liver disease
* History or other evidence of a medical condition associated with chronic liver disease other than viral hepatitis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- China (7):
  - Changsha
  - Chengdu
  - Fuzhou
  - Guangzhou
  - Hangzhou
  - Wuhan
  - Xi'an

REFERENCES:
- [Derived] Yan W, Wu D, Wang X, Chen T, Lai Q, Zheng Q, Jiang J, Hou J, Han M, Ning Q. Upregulation of NKG2C+ natural killer cells, TLR-2 expression on monocytes and downregulation of regulatory T-cells influence PEG-IFN treatment efficacy in entecavir-suppressed patients with CHB. Antivir Ther. 2015;20(6):591-602. doi: 10.3851/IMP2953. Epub 2015 Mar 27. PMID 25814467
- [Derived] Ning Q, Han M, Sun Y, Jiang J, Tan D, Hou J, Tang H, Sheng J, Zhao M. Switching from entecavir to PegIFN alfa-2a in patients with HBeAg-positive chronic hepatitis B: a randomised open-label trial (OSST trial). J Hepatol. 2014 Oct;61(4):777-84. doi: 10.1016/j.jhep.2014.05.044. Epub 2014 Jun 7. PMID 24915612

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 332 participants were enrolled in this study conducted from 28 April 2009 to 23 December 2011 at seven centers in China.
Pre-assignment Details: Of 332 participants, 200 were randomized, out of which 97 participants were assigned to Peginterferon alfa-2a + entecavir and 100 were assigned to entecavir, and three participants did not take any study drug.
Period: Overall Study
Arm/Group | Peginterferon Alfa-2a + Entecavir | Entecavir
Started | 97 | 100
Completed | 82 | 93
Not Completed | 15 | 7
Not completed — HBeAb positive at Baseline | 3 | 2
Not completed — Lost to Follow-up | 2 | 3
Not completed — Adverse Event | 8 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Others | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized subjects who had baseline evaluations and at least one efficacy evaluation.
Groups:
- Peginterferon Alfa-2a + Entecavir: Participants received peginterferon alfa-2a180 mcg subcutaneously once weekly for 48 weeks, plus entecavir 0.5 mg orally once daily for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Peginterferon Alfa-2a + Entecavir | Entecavir | Total
Number analyzed (Participants) | 94 | 98 | 192
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.38 (8.25) | 33.28 (8.95) | 33.3 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 13 | 32
  Male | 75 | 85 | 160

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Hepatitis B Envelope Antigen Seroconversion at Week 48
Description: Hepatitis B envelope Antigen (HBeAg) seroconversion was defined as the absence of HBeAg and the presence of antibody to Hepatitis B envelope antigen (anti-HBe).
Time Frame: At Week 48
Population: Full analysis set included all patients who were randomized and received at least one dose of the study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Peginterferon Alfa-2a + Entecavir | Entecavir
Number analyzed (Participants) | 94 | 98
Percentage of participants | 14.89 [8.39 to 23.72] | 6.12 [2.28 to 12.85]

2. Secondary Outcome: Percentage of Participants With Loss of Hepatitis B Envelope Antigen at Week 48
Description: Loss of Hepatitis B Envelope Antigen (HBeAg) is defined as the absence of HBeAg.
Time Frame: At Week 48
Population: Full analysis set included all patients who were randomized and received at least one dose of the study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Peginterferon Alfa-2a + Entecavir | Entecavir
Number analyzed (Participants) | 94 | 98
Percentage of participants | 62.77 [52.18 to 72.52] | 60.20 [49.82 to 69.96]

3. Secondary Outcome: Percentage of Participants With Hepatitis B Virus - Deoxyribonucleic Acid <1000 Copies/ Millilitre at Week 48
Description: Blood was collected for Hepatitis B Virus - Deoxyribonucleic Acid (HBV -DNA) and was analysed at the central laboratories using the Roche approved polymerase chain reaction (PCR) methodology at Week 48. Percentage of participants with HBV-DNA < 1000 copies/mL was reported.
Time Frame: At Week 48
Population: Full analysis set included all patients who were randomized and received at least one dose of the study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Peginterferon Alfa-2a + Entecavir | Entecavir
Number analyzed (Participants) | 94 | 98
Percentage of participants | 62.77 [52.18 to 72.52] | 91.84 [84.55 to 96.41]

4. Secondary Outcome: Percentage of Participants With Hepatitis B Surface Antigen Loss at Week 48
Description: Loss of Hepatitis B Surface Antigen (HBsAg) was defined as change of detectable HBsAg from positive to negative.
Time Frame: At Week 48
Population: Full analysis set included all patients who were randomized and received at least one dose of the study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Peginterferon Alfa-2a + Entecavir | Entecavir
Number analyzed (Participants) | 94 | 98
Percentage of participants | 8.51 [3.75 to 16.08] | 0 [0 to 3.69]

5. Secondary Outcome: Percentage of Participants With Hepatitis B Surface Antigen Seroconversion at Week 48
Description: Hepatitis B Surface Antigen (HBsAg) seroconversion was defined as loss of HBsAg and presence of anti-HBs .(antibody to Hepatitis B surface antigen)
Time Frame: At Week 48
Population: Full analysis set included all patients who were randomized and received at least one dose of the study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Peginterferon Alfa-2a + Entecavir | Entecavir
Number analyzed (Participants) | 94 | 98
Percentage of participants | 4.26 [1.17 to 10.54] | 0 [0 to 3.69]

6. Secondary Outcome: Percentage of Participants With Normalized Alanine Aminotransferase at Week 48
Description: Normalized Alanine Aminotransferase (ALT) is defined as having a baseline ALT value > upper limit of normal (ULN), and a decrease in ALT value to ≤ ULN at the given time point.
Time Frame: At Week 48
Population: Full analysis set included all patients who were randomized and received at least one dose of the study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Peginterferon Alfa-2a + Entecavir | Entecavir
Number analyzed (Participants) | 94 | 98
Percentage of participants | 51.06 [40.54 to 61.52] | 85.71 [77.19 to 91.96]

7. Secondary Outcome: Quantitative Change in Mean Hepatitis B Envelope Antigen Over Time
Description: Quantitative hepatitis B envelope antigen (HBeAg) results were analyzed in central lab. Values that were less than lower limit of quantification (LLOQ) had been replaced by LLOQ when analyzed, e.g. <1000 was replaced by 1000 and <0.2 was replaced by 0.2. Quantitative HBeAg value unit was calculated using 'Paul Ehrlich Institute units per millilitre' (PEIU/ml). Change in HBeAg was analysed at Weeks 0, 8, 12, 24, 36, and 48.
Time Frame: Up to Week 48
Population: Full analysis set included all patients who were randomized and received at least one dose of the study drug. Maximum participants available at particular time point were analysed.
Measure: Mean (Standard Deviation); unit: PEIU/ml)
Arm/Group | Peginterferon Alfa-2a + Entecavir | Entecavir
Number analyzed (Participants) | 94 | 97
PEIU/ml)
  At Week 0; n= 93, 95 | 8.33 (18.76) | 5.66 (10.33)
  At Week 8; n= 93, 97 | 4.76 (11.63) | 5.85 (12.55)
  At Week 12; n= 94, 97 | 3.83 (10.57) | 5.00 (10.56)
  At Week 24; n= 91, 97 | 2.28 (5.81) | 4.76 (11.40)
  At Week 36; n= 88, 94 | 3.58 (16.66) | 4.52 (10.10)
  At Week 48; n= 85, 92 | 13.23 (93.02) | 4.07 (9.15)

8. Secondary Outcome: Quantitative Change in Mean Hepatitis B Surface Antigen Change Over Time
Description: Quantitative Hepatitis B Surface Antigen (HBsAg) results were analyzed in central lab. Values that were less than LLOQ had been replaced by LLOQ when analyzed, e.g. <1000 was replaced by 1000 and <0.2 was replaced by 0.2. Quantitative HBsAg calculated using 'International Units Per Millilitre' (IU/mL). Change in HBsAg was analysed at Weeks 0, 8, 12, 24, 36, and 48.
Time Frame: Up to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: IU/ml
Arm/Group | Peginterferon Alfa-2a + Entecavir | Entecavir
Number analyzed (Participants) | 94 | 97
IU/ml
  At Week 0; n= 93, 95 | 3737.84 (4617.19) | 3241.06 (3592.60)
  At Week 8; n= 93, 97 | 3603.56 (4553.66) | 3050.79 (3313.12)
  At Week 12; n= 94, 97 | 3041.86 (3782.70) | 3037.82 (3498.73)
  At Week 24; n= 91, 97 | 2280.60 (3429.61) | 2895.25 (3336.91)
  At Week 36; n= 88, 94 | 2097.89 (3458.84) | 2699.18 (2964.25)
  At Week 48; n= 85, 92 | 1886.02 (2627.33) | 2672.71 (3065.97)

9. Secondary Outcome: Number of Participants With Incidence of Adverse Events and Serious Adverse Events
Description: An adverse event (AE) was defined as any untoward medical occurrence that occurred during the course of the trial after study treatment had started. An adverse event was therefore any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. A Serious Adverse Events (SAE) is any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity, and congenital anomaly/birth defect.
Time Frame: Up to Week 48
Population: Safety set (SS) included all the participants who received at least 1 dose of study drug and who had at least undergone safety assessment once, regardless of whether the patients withdrew from the study or not.
Measure: Number; unit: Participants
Arm/Group | Peginterferon Alfa-2a + Entecavir | Entecavir
Number analyzed (Participants) | 97 | 100
Participants
  Non serious AE | 65 | 5
  Serious AE | 6 | 0
  AE | 67 | 5

10. Secondary Outcome: Number of Participants With Laboratory Abnormalities Which Were Captured as an Adverse Event
Description: Participants with clinically significant laboratory abnormalities which were captured as an AE (at the >=5% threshold) were presented.
Time Frame: Up to Week 48
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | Peginterferon Alfa-2a + Entecavir | Entecavir
Number analyzed (Participants) | 97 | 100
Participants
  Haemoglobin decreased | 6 | 0
  Aspartate aminotransferase increased | 8 | 0
  Alanine aminotransferase increased | 9 | 0
  Platelet count decreased | 42 | 0
  Neutrophil count decreased | 53 | 0
  White blood cell count decreased | 59 | 0

ADVERSE EVENTS:
Time Frame: Up to Week 48
Description: Serious adverse events and non-serious adverse events are reported in Safety Analysis Set, which consists of all participants who received at least one dose of study medication and had a safety assessment performed post baseline.
Arm/Group | Peginterferon Alfa-2a + Entecavir | Entecavir
Serious Adverse Events (participants affected / at risk) | 6/97 | 0/100
Other Adverse Events (participants affected / at risk) | 65/97 | 5/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peginterferon Alfa-2a + Entecavir (N=97) | Entecavir (N=100)
Hypothyroidism (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 0
Viral myocarditis (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peginterferon Alfa-2a + Entecavir (N=97) | Entecavir (N=100)
Haemoglobin decreased (Investigations) | 6 | 0
Aspartate aminotransferase increased (Investigations) | 8 | 0
Alanine aminotransferase increased (Investigations) | 9 | 0
Platelet count decreased (Investigations) | 42 | 0
Neutrophil count decreased (Investigations) | 53 | 0
White blood cell count decreased (Investigations) | 59 | 0
Pyrexia (General disorders) | 15 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 0
Erythropenia (Blood and lymphatic system disorders) | 5 | 0
Red blood cells urine positive (Investigations) | 0 | 1
Ultrasound liver abnormal (Investigations) | 0 | 1
Blood thyroid stimulating hormone decreased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Protein urine present (Investigations) | 1 | 0
Thyroxine increased (Investigations) | 1 | 0
Tri-iodothyronine increased (Investigations) | 1 | 0
White blood cells urine positive (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 2 | 0
Weight decreased (Investigations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Pharyngitis (Infections and infestations) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Influenza like illness (General disorders) | 3 | 0
Conjunctivitis (Eye disorders) | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 3 | 0
Marasmus (Metabolism and nutrition disorders) | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 4 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Headache (Nervous system disorders) | 4 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.